CLINICAL TRIAL: NCT00001270
Title: Feasibility Study of Interleukin 1-Alpha With Ifosfamide, CBDCA, and Etoposide With Autologous Bone Marrow Transplant in Metastatic Carcinoma and Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 910156; 91-C-0156
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Breast Neoplasms; Lymphoma; Neoplasm Metastasis; Testicular Neoplasms
Keywords: Chemotherapy; High Dose; Protection
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Neoplasm Metastasis; Testicular Neoplasms | interventions — Interleukin-1

INTERVENTIONS:
Drug: interleukin-1

SUMMARY:
This is a phase I/II study of interleukin-1, G-CSF and high dose ICE chemotherapy with autologous bone marrow transplant in patients with relapsed breast, testicular and lymphoid cancers. The initial goal of this study was to define the toxicity of interleukin-1 administered for 7 days prior to ICE chemotherapy. A total of 22 patients have been treated with IL-1 and ICE and results showed a more rapid engraftment (4.5 days) with IL-1. A second cohort of 18 patients also received G-CSF and engraftment was further shortened in some subgroups. Overall, the median time to engraftment was 16 days with both IL-1 and G-CSF. Accrual will continue to further define the toxicity and efficacy of this regimen.

DETAILED DESCRIPTION:
This is a phase I/II study of interleukin-1, G-CSF and high dose ICE chemotherapy with autologous bone marrow transplant in patients with relapsed breast, testicular and lymphoid cancers. The initial goal of this study was to define the toxicity of interleukin-1 administered for 7 days prior to ICE chemotherapy. A total of 22 patients have been treated with IL-1 and ICE and results showed a more rapid engraftment (4.5 days) with IL-1. A second cohort of 18 patients also received G-CSF and engraftment was further shortened in some subgroups. Overall, the median time to engraftment was 16 days with both IL-1 and G-CSF. Accrual will continue to further define the toxicity and efficacy of this regimen.

ELIGIBILITY:
A history of pathologically documented (clinical documentation may be acceptable at relapse):

Breast cancer: metastatic or locally advanced (Stage III/IV) with stable minimal (less than or equal to 2 cm) residual disease after 2 cycles of appropriate combination chemotherapy may start BMT.

Non-Hodgkin's lymphomas: all stages of relapsed or induction failure (FSC, FM, FL, DSC, DL, DM, DIDL, IBL, LBL, SNC) after appropriate chemotherapy.

Hodgkin's lymphomas: all stages of chemotherapy induction failures, first relapse less than or equal to 1 year from chemotherapy induced remission, first relapse greater than 1 year from chemotherapy induced remission if there is extranodal involvement at relapse, greater than or equal to 2 relapses (one may be after radiation) following appropriate combination chemotherapy, or relapse at any time from radiation therapy with stage IIB, IIIB, IV A/B.

Testicular cancer: all stages of relapsed or induction failure following appropriate combination chemotherapy.

No evidence of central nervous system cancer.

Patients must be between 18 and 65 years old.

Normal cardiac function: no history of angina pectoris, myocardial infarction, congestive heart failure or ejection fraction less than 40 percent.

Creatinine clearance greater than or equal to 45 cc/min/m(2), bilirubin less than or equal to 1.5, SGOT less than or equal to 2x normal, and normal PT, PTT and calcium.

Negative HIV serology and hepatitis B surface antigen.

Adequate pulmonary function (PFTs are only obtained in patients with clinical evidence of pulmonary dysfunction): DLCO greater than 50 percent, compensated for Hgb, FEV 1 greater than 55 percent and PO2 greater than 60.

Negative bilateral bone marrow biopsies prior to bone marrow harvest.

No evidence of metastatic disease to the pelvis on plain film or bone scan.

Karnofsky performance status greater than or equal to 70 and a life expectancy greater than or equal to 60 days.

No evidence of pregnancy or risk of pregnancy at the time of transplantation in women.

Ability to give informed consent.

Good psychiatric and medical risk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85
Dates: Start 1991-06; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Jagannath S, Dicke KA, Armitage JO, Cabanillas FF, Horwitz LJ, Vellekoop L, Zander AR, Spitzer G. High-dose cyclophosphamide, carmustine, and etoposide and autologous bone marrow transplantation for relapsed Hodgkin's disease. Ann Intern Med. 1986 Feb;104(2):163-8. doi: 10.7326/0003-4819-104-2-163. PMID 3511811
- [Background] Neta R, Oppenheim JJ. Cytokines in therapy of radiation injury. Blood. 1988 Sep;72(3):1093-5. PMID 2458148